CLINICAL TRIAL: NCT06178783
Title: A Phase 1, Double-blind, Randomized, Single-center Study to Assess the Palatability and Acceptability of Different Brensocatib Oral Liquid Formulations in Healthy Subjects
Brief Title: A Study of the Palatability and Acceptability of Different Brensocatib Oral Liquid Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INS1007-107; 8521537 (Other: Fortrea)
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — brensocatib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Brensocatib Treatment Sequence ADBC (Experimental): Participants will taste and expectorate Dose 1 of each brensocatib formulation across the 4 treatment administrations (Treatments A, B, C, and D), orally on Day 1 in the sequence ADBC.
  Interventions: Drug: Brensocatib
- Brensocatib Treatment Sequence BACD (Experimental): Participants will taste and expectorate Dose 1 of each brensocatib formulation across the 4 treatment administrations (Treatments A, B, C, and D), orally on Day 1 in the sequence BACD.
  Interventions: Drug: Brensocatib
- Brensocatib Treatment Sequence CBDA (Experimental): Participants will taste and expectorate Dose 1 of each brensocatib formulation across the 4 treatment administrations (Treatments A, B, C, and D), orally on Day 1 in the sequence CBDA.
  Interventions: Drug: Brensocatib
- Brensocatib Treatment Sequence DCAB (Experimental): Participants will taste and expectorate Dose 1 of each brensocatib formulation across the 4 treatment administrations (Treatments A, B, C, and D), orally on Day 1 in the sequence DCAB.
  Interventions: Drug: Brensocatib

INTERVENTIONS:
Drug: Brensocatib — Brensocatib oral solutions will be expectorated following the tasting.
  Other Names: INS1007; AZD7986

SUMMARY:
The primary purpose of this study is to assess the palatability and compare acceptability of brensocatib oral solutions.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kilogram per meter square (kg/m^2), inclusive, and a body weight of ≥50 kilograms (kg) at screening.
* In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG), vital signs measurements, clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable), and physical examination at screening and/or Day 1, as assessed by the investigator (or designee).
* Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.

Exclusion Criteria:

* Positive hepatitis panel and/or positive human immunodeficiency virus test.
* The participant has a mouth pathology including, but not limited to, pain, ulcer, edema, mucosal erosion, and/or (dental) abscesses, or receives treatment for oral pathologies or oral treatment for any disease.
* The participant is unable to taste and smell normally, to his/her own opinion, at any time throughout the study duration Participants who have an impaired sense of taste and/or smell due to any conditions like common cold or sinusitis are not eligible to take part or continue the study.
* Administration of a vaccine in the past 14 days prior to Day 1.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 60 days or 5 half-lives of that drug prior to Day 1, whichever is longer.
* History of alcoholism or drug/chemical abuse within 2 years prior to Day 1.
* Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
* Poor peripheral venous access.

Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants With High Acceptability to Each Brensocatib Formulation Based on Palatability Assessments Measured by the 9-point Hedonic Scale | Day 1

SECONDARY OUTCOMES:
Number of Participants who Experienced at Least one Adverse Event (AE) | Up to Day 4
  Determination of the tolerability of brensocatib oral solutions in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- USA001, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No